CLINICAL TRIAL: NCT06988228
Title: The Effects of 15% Dextrose Solution on Pain and Range of Motion in the Hemiplegic Shoulder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, ayseyildirim, principal investigator, Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SBUSAH-GETAT 2024-057; SBUSAH-GETAT (Other: 2024-057)
Record Dates: First submitted 2025-05-17; First posted 2025-05-23 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-05

CONDITIONS: Hemiplegic Shoulder Pain; Stroke
Keywords: %15 prolotherapy; %15 dextrose injection; hemiplegic shoulder pain; post-stroke rehabilitation; fugl-meyer; barthel ındex
MeSH Terms: conditions — Stroke | interventions — Glucose

STUDY DESIGN:
Intervention Model Description: The study includes two parallel groups. Both receive conventional exercise therapy. The intervention group receives three sessions of 15% dextrose solution injections, and the control group receives three sessions of isotonic saline solution injections, administered at two-week intervals.
Who Masked: Participant
Masking Description: This is a single-blinded study. Participants are blinded to the type of solution (dextrose or isotonic saline) administered during the injections.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Participants in this group will receive three sessions of 15% dextrose solution injections at two-week intervals, in addition to conventional exercise therapy.
  Interventions: Biological: 15% Dextrose Injection
- control group (Placebo Comparator): Participants in this group will receive three sessions of isotonic saline solution injections at two-week intervals, in addition to conventional exercise therapy.
  Interventions: Other: izotonic saline injection

INTERVENTIONS:
Biological: 15% Dextrose Injection — 15% dextrose solution will be administered by injection in three sessions at two-week intervals. It will be applied in combination with conventional exercise therapy.
  Arms: intervention group
Other: izotonic saline injection — Participants will receive isotonic saline solution injections in three sessions at two-week intervals, as a placebo comparator to the 15% dextrose injections. All participants will also receive conventional exercise therapy.
  Arms: control group

SUMMARY:
This study aims to investigate the effects of 15% dextrose solution on pain and range of motion in patients aged 40 to 75 years who have experienced a stroke and suffering from hemiplegic shoulder pain

DETAILED DESCRIPTION:
This randomized, controlled, single-blinded clinical trial aims to evaluate the effects of 15% dextrose solution on pain and shoulder range of motion in patients with hemiplegic shoulder pain following a stroke. A total of 40 participants aged 40 to 75 years will be enrolled and randomly assigned into two groups of equal size.

Both groups will receive conventional exercise therapy. In addition, the intervention group will receive three sessions of 15% dextrose solution injections administered at two-week intervals, whereas the control group will receive three sessions of isotonic saline solution injections on the same schedule.

Assessments will be conducted at baseline, one month after the final injection, and three months after the final injection. The primary outcome measure is the change in pain intensity. Secondary outcome measures include goniometric range of motion (ROM) evaluation, Visual Analog Scale (VAS), Barthel Index for functional independence, and the shoulder section of the Fugl-Meyer Upper Extremity Motor Assessment Scale(Shoulder subsection).

This study aims to determine whether 15% dextrose prolotherapy offers superior clinical outcomes in reducing pain and improving functional status compared to isotonic saline injection when combined with a standard exercise program.

ELIGIBILITY:
Inclusion Criteria:

Patients aged between 40 and 75 years

History of stroke

Brunnstrom stage 2 or higher in the upper extremity

Provided written informed consent and agreed to participate in the study

Exclusion Criteria:

History of any prior injection therapy to the shoulder region

Previous radiotherapy or surgery involving the shoulder

Pre-stroke shoulder pain

History of shoulder surgery

History of inflammatory joint disease

Presence of neuromuscular disorders

Full-thickness rotator cuff tear

Patients with aphasia or severe cognitive impairment

Presence of pectoral muscle spasticity

Active malignancy with acute inflammation at the treatment site

Known coagulation disorder with INR ≥ 4

Presence of vascular conditions such as deep vein thrombosis, phlebitis, varicose veins, or arterial disease in the affected limb

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-12-24 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Pain intensity measured by Visual Analog Scale (VAS, 0-10 cm; higher scores = worse pain) | Baseline, 1 month after last injection, 3 months after last injection
  Pain intensity will be assessed using the Visual Analog Scale (VAS), a 10-centimeter scale ranging from 0 (no pain) to 10 (worst imaginable pain). Higher scores indicate worse outcomes (greater pain intensity). Pain will be evaluated in three different conditions: at rest, after exercise, and during daily activities. Participants will rate their pain separately for each condition. The change in VAS scores from baseline to 1 month and 3 months after the final injection will be evaluated.

SECONDARY OUTCOMES:
Shoulder Range of Motion (ROM) measured using a standard goniometer (abduction and flexion, degrees) | Baseline, 1 month after last injection, 3 months after last injection
  Shoulder joint mobility will be assessed using a standard manual goniometer. Active range of motion will be measured in degrees for shoulder abduction and flexion only. Measurements will be taken on the affected (hemiplegic) side with the participant in a seated position. Higher values indicate better outcomes (greater joint mobility). Changes from baseline to 1 month and 3 months after the final injection will be evaluated.
Barthel Index Score (range 0-100; higher scores = better functional independence) | Baseline, 1 month after last injection, 3 months after last injection
  Functional independence in activities of daily living (ADLs) will be assessed using the Barthel Index, a standardized scale that evaluates a person's ability to perform 10 basic self-care and mobility tasks. The total score ranges from 0 to 100, with higher scores indicating better functional status and greater independence. The change in Barthel Index scores from baseline to 1 month and 3 months after the final injection will be analyzed.
Fugl-Meyer Assessment - Upper Extremity (Shoulder Subsection) Score (range 0-40; higher scores = better motor function) | Baseline, 1 month after last injection, 3 months after last injection
  Motor function of the affected upper limb will be assessed using the shoulder subsection of the Fugl-Meyer Assessment of Upper Extremity (FMA-UE). This subsection evaluates reflex activity, voluntary movement within and outside synergy patterns, and coordination of shoulder and elbow movements. The score ranges from 0 to 40, with higher scores indicating better motor recovery. Changes from baseline to 1 month and 3 months after the final injection will be analyzed.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Physical Medicine and Rehabilitation Training and Research Hospital, Istanbul, bahçelievler, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be available upon reasonable request from qualified researchers after the publication of study results. Data sharing will require approval by the principal investigator and compliance with ethical guidelines.
Supporting Information: Study Protocol, SAP
Time Frame: De-identified IPD and supporting information will be available 6 months after publication of the primary results and will remain accessible for up to 3 years.
Access Criteria: Qualified researchers may request access to the IPD and supporting documents. Requests will be reviewed and approved by the principal investigator. A data use agreement and adherence to ethical standards will be required.

REFERENCES:
- [Background] Coskun Benlidayi I, Basaran S. Hemiplegic shoulder pain: a common clinical consequence of stroke. Pract Neurol. 2014 Apr;14(2):88-91. doi: 10.1136/practneurol-2013-000606. Epub 2013 Aug 12. PMID 23940374
- [Background] Hauser RA, Lackner JB, Steilen-Matias D, Harris DK. A Systematic Review of Dextrose Prolotherapy for Chronic Musculoskeletal Pain. Clin Med Insights Arthritis Musculoskelet Disord. 2016 Jul 7;9:139-59. doi: 10.4137/CMAMD.S39160. eCollection 2016. PMID 27429562
- [Background] Thor JA, Mohamed Hanapi NH, Halil H, Suhaimi A. Perineural Injection Therapy in the Management of Complex Regional Pain Syndrome: A Sweet Solution to Pain. Pain Med. 2017 Oct 1;18(10):2041-2045. doi: 10.1093/pm/pnx063. No abstract available. PMID 28460075
- [Background] Kumar P. Hemiplegic shoulder pain in people with stroke: present and the future. Pain Manag. 2019 Mar 1;9(2):107-110. doi: 10.2217/pmt-2018-0075. Epub 2019 Jan 25. No abstract available. PMID 30681020
- [Background] Mansiz-Kaplan B, Nacir B, Pervane-Vural S, Tosun-Meric O, Duyur-Cakit B, Genc H. Effect of Perineural Dextrose Injection on Ulnar Neuropathy at the Elbow: A Randomized, Controlled, Double-Blind Study. Arch Phys Med Rehabil. 2022 Nov;103(11):2085-2091. doi: 10.1016/j.apmr.2022.04.013. Epub 2022 Jun 9. PMID 35690093